CLINICAL TRIAL: NCT04662281
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of LX9211 in the Treatment of Postherpetic Neuralgia (RELIEF-PHN1)
Brief Title: Efficacy and Safety of LX9211 in Participants With Postherpetic Neuralgia
Acronym: RELIEF-PHN1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX9211.1-202-PHN; 2020-004639-26 (EudraCT Number)
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Following a 2-week Single-blind Run-in period, participants will receive a single loading dose of matching-placebo to LX9211 tablet, orally, on Day 1 and maintenance doses, orally, once daily from Day 2 to Week 6.
  Interventions: Drug: Placebo
- LX9211 (Experimental): Following a 2-week Single-blind Run-in period, participants will receive a single loading dose of 200 milligrams (mg) tablet, orally, on Day 1 and maintenance doses of 20 mg, orally, once daily from Day 2 to Week 6.
  Interventions: Drug: LX9211

INTERVENTIONS:
Drug: Placebo — LX9211 matching-placebo, tablets will be administered orally.
  Arms: Placebo
Drug: LX9211 — LX9211, 200 mg, tablets will be administered orally.
  Arms: LX9211

SUMMARY:
Evaluation of the efficacy of LX9211 compared to placebo in reducing pain related to postherpetic neuralgia over an 11 week assessment period.

ELIGIBILITY:
Inclusion Criteria:

* Participant has given written informed consent to participate in the study in accordance with local regulations
* Adult male and female participants ≥18 years of age at the time of screening
* PHN pain that is present for ≥3 months after healing of herpes zoster skin rash affecting a single dermatome (Participants with more than 1 involved dermatome may also be included, provided the affected dermatomes are contiguous)
* Moderate to severe pain as confirmed by average pain score using scores recorded in the pain diary in the 14 days prior to randomization

Exclusion Criteria:

* Presence of other painful conditions that may confound assessment or self-evaluation of PHN
* History of major depressive episode, active, significant psychiatric disorders
* History of clinically significant drug or alcohol use disorder
* PHN affecting the face
* Use of opioid medications for management of PHN within the 2 months prior to Screening Visit
* Use of Non-steroidal anti-inflammatory drugs (NSAIDs) for the specific treatment of PHN pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Average Daily Pain Score (ADPS) | Day 1 to Week 6
  The change from Baseline (Week 2) to Week 6 in Average Daily Pain Score (ADPS), based on the 11-point numerical rating scale (0 [No Pain] to 10 [Pain as bad as you can imagine])

SECONDARY OUTCOMES:
≥30 percent reduction in pain intensity | Day 1 to Week 6
  Proportion of patients with ≥30% reduction in pain intensity
≥50 percent reduction in pain intensity | Day 1 to Week 6
  Proportion of patients with ≥50% reduction in pain intensity
Safety: number of AEs reported | Day 1 to Week 6
  Number of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Suma Gopinathan, PhD, Study Director — Lexicon Pharmaceuticals
Locations (31):
- United States (21):
  - Lexicon Investigational Site, Scottsdale, Arizona
  - Lexicon Investigational Site, Tucson, Arizona
  - Lexicon Investigational Site, Greenbrae, California
  - Lexicon Investigational Site, Brandon, Florida
  - Lexicon Investigational Site (113), Miami, Florida
  - Lexicon Investigational Site, Miami, Florida
  - Lexicon Investigational Site, Ormond Beach, Florida
  - Lexicon Investigational Site, Winter Park, Florida
  - Lexicon Investigational Site (147), Marietta, Georgia
  - Lexicon Investigational Site, Flossmoor, Illinois
  - Lexicon Investigational Site, Wauconda, Illinois
  - Lexicon Investigational Site, Boston, Massachusetts
  - Lexicon Investigational Site, Canton, Michigan
  - Lexicon Investigational Site, Hazelwood, Missouri
  - Lexicon Investigational Site, Albuquerque, New Mexico
  - Lexicon Investigational Site (148), Cary, North Carolina
  - Lexicon Investigational Site, Jenkintown, Pennsylvania
  - Lexicon Investigational Site, Baytown, Texas
  - Lexicon Investigational Site, Victoria, Texas
  - Lexicon Investigational Site, Salt Lake City, Utah
  - Lexicon Investigational Site, Kenosha, Wisconsin
- Czechia (6):
  - Lexicon Investigational Site (138), Choceň
  - Lexicon Investigational Site (140), Pardubice
  - Lexicon Investigational Site (136), Prague
  - Lexicon Investigational Site (137), Prague
  - Lexicon Investigational Site (141), Prague
  - Lexicon Investigational Site (135), Prague
- Poland (4):
  - Lexicon Investigational Site (128), Katowice
  - Lexicon Investigational Site (130), Katowice
  - Lexicon Investigational Site (134), Lublin
  - Lexicon Investigational Site (133), Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Luo G, Chen L, Kostich WA, Hamman B, Allen J, Easton A, Bourin C, Gulianello M, Lippy J, Nara S, Maishal TK, Thiyagarajan K, Jalagam P, Pattipati SN, Dandapani K, Dokania M, Vattikundala P, Sharma V, Elavazhagan S, Verma MK, Das ML, Wagh S, Balakrishnan A, Johnson BM, Santone KS, Thalody G, Denton R, Saminathan H, Holenarsipur VK, Kumar A, Rao A, Putlur SP, Sarvasiddhi SK, Shankar G, Louis JV, Ramarao M, Conway CM, Li YW, Pieschl R, Tian Y, Hong Y, Ditta J, Mathur A, Li J, Smith D, Pawluczyk J, Sun D, Yip S, Wu DR, Vetrichelvan M, Gupta A, Wilson A, Gopinathan S, Wason S, Bristow L, Albright CF, Bronson JJ, Macor JE, Dzierba CD. Discovery of (S)-1-((2',6-Bis(difluoromethyl)-[2,4'-bipyridin]-5-yl)oxy)-2,4-dimethylpentan-2-amine (BMS-986176/LX-9211): A Highly Selective, CNS Penetrable, and Orally Active Adaptor Protein-2 Associated Kinase 1 Inhibitor in Clinical Trials for the Treatment of Neuropathic Pain. J Med Chem. 2022 Mar 24;65(6):4457-4480. doi: 10.1021/acs.jmedchem.1c02131. Epub 2022 Mar 8. PMID 35257579